CLINICAL TRIAL: NCT00727350
Title: Phase II Protocol for Primary Fractionated Stereotactic Body Radiation Therapy for Stage T1 - T3N0 Non Small Cell Lung Carcinoma.
Brief Title: Protocol for Primary Fractionated Stereotactic Body Radiation Therapy for Stage T1 - T3N0 Non Small Cell Lung Carcinoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AZ-VUB (Other)
Responsible Party: Samuel Bral, AZ-VUB
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBRT-NSCLC
Record Dates: First submitted 2008-07-31; First posted 2008-08-04 (Estimated); Last update posted 2008-08-04 (Estimated); Status verified 2008-08

CONDITIONS: Non Small Cell Lung Carcinoma
Keywords: NSCLC; Novalis; Stereotactic; SBRT; T1, T2 or T3NO NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): For centrally located T1 and T2 lesions 4 x 15 Gy over 2 weeks will be delivered. Lesions located peripherally will be treated with 3 x 20 Gy, also delivered within 2 weeks. For both schedules, there should be a minimum of 40 hours and a maximum of 8 days between 2 separate fractions. There should be a maximum of 2 fractions per week.
  Interventions: Radiation: Fractionated stereotactic body radiation therapy

INTERVENTIONS:
Radiation: Fractionated stereotactic body radiation therapy — For centrally located T1 and T2 lesions 4 x 15 Gy over 2 weeks will be delivered. Lesions located peripherally will be treated with 3 x 20 Gy, also delivered within 2 weeks. For both schedules, there should be a minimum of 40 hours and a maximum of 8 days between 2 separate fractions. There should be a maximum of 2 fractions per week.

SUMMARY:
The study population will exist of patients with a histological diagnosis of NSCLC, stage T1, T2 or T3NO who are not fit for or who refuse surgery. A prospective data analysis will be performed on tumor response, potential acute and late toxicity and survival. A radiotherapy dose of 4x15Gy or 3x 20Gy will be given over 2 weeks with dynamic 3D-conformal arc therapy (Novalis TM)

ELIGIBILITY:
Inclusion Criteria:

1. Stage T1,T2,T3N0M0 NSCLC, histological confirmation either by biopsy or cytology
2. Maximal tumor diameter of 6 cm
3. Only T3 lesions based upon thoracic wall involvement
4. Informed consent is required
5. Life expectancy of at least 6 months
6. Age > 18 y.
7. Karnofsky score ≥ 70 or ECOG score ≤ 1
8. Inoperable patients or patients refusing surgery
9. Patients with measurable lesion (according to RECIST criteria)

Exclusion Criteria:

1. Diagnosis of small cell lung cancer
2. Lymph node involvement
3. Prior radiotherapy or chemotherapy for lung cancer
4. Pregnant or lactating women
5. Known allergy for CT contrast
6. No FDG-PET
7. Mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study.
8. Patient unlikely to comply with protocol, i.e., uncooperative attitude, inability to return for follow-up visits, extreme degradation of lung function tests and patients not likely to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2007-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To monitor potential acute and late toxicity in patients with stage T1,T2,T3N0 non small cell lung carcinoma (NSCLC), treated with primary stereotactic body radiation therapy (SBRT). | Every 3 months for the first 2 years. From 3 to 5 years every 6 months. After 5 years follow-up will happen yearly.

SECONDARY OUTCOMES:
Local control at 2 years. Overall survival, local progression free survival, disease free survival, time to progression and local,regional or disseminated recurrence.Quality of life. Internal and Intra-fractional tumor motion. Biopsy samples. | Every 3 months for the first 2 years. From 3 to 5 years every 6 months. After 5 years follow-up will happen yearly.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

REFERENCES:
- [Derived] Bral S, Gevaert T, Linthout N, Versmessen H, Collen C, Engels B, Verdries D, Everaert H, Christian N, De Ridder M, Storme G. Prospective, risk-adapted strategy of stereotactic body radiotherapy for early-stage non-small-cell lung cancer: results of a Phase II trial. Int J Radiat Oncol Biol Phys. 2011 Aug 1;80(5):1343-9. doi: 10.1016/j.ijrobp.2010.04.056. Epub 2010 Aug 12. PMID 20708849